CLINICAL TRIAL: NCT01844583
Title: Study of the Effect of Esomeprazole or Rifampin on the Pharmacokinetics of Alisertib and Evaluation of the Effect of Alisertib on the QTc Interval in Patients With Advanced Solid Tumors or Lymphomas
Brief Title: Safety, Tolerability and Pharmacokinetic (PK) of Concomitant Esomeprazole and Rifampin, and QT Study on Single and Multiple-doses of Alisertib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C14015
Record Dates: First submitted 2013-04-29; First posted 2013-05-01 (Estimated); Results first posted 2019-03-25 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2018-12

CONDITIONS: Solid Tumors; Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — MLN 8237; Esomeprazole; Rifampin

ARMS (2):
- Esomeprazole 40 mg + Alisertib 50 mg (Experimental): Alisertib 50 mg, tablets, orally, once on Day 1, followed by twice daily on Days 4 to 10, followed by a 14-day rest period in Cycle 1.
  Esomeprazole, 40 mg, delayed-release capsules, orally, once daily on Days 1 to 10 plus alisertib, 50 mg, tablets, orally, once on Day 8, followed by twice daily on Days 11 to 17, followed by a 14-day rest period in Cycle 2.
  Alisertib 50 mg, tablets, orally, twice daily on Days 1 to 7 beginning with Cycle 3 (21-day cycles) to the end of study (Up to 15 Cycles).
  Interventions: Drug: Alisertib; Drug: Esomeprazole
- Rifampin 600 mg + Alisertib 50 mg (Experimental): Alisertib 50 mg, tablets, orally, once on Day 1, followed by twice daily on Days 4 to 10, followed by a 14-day rest period in Cycle 1.
  Rifampin 600 mg, capsules, orally, once daily on Days 1 to 10 in Cycle 2 plus alisertib, 50 mg, tablets, orally, once on Day 8, followed by twice daily on Days 11 to 17, followed by a 14-day rest period in Cycle 2.
  Alisertib 50 mg, tablets, orally, twice daily on Days 1 to 7 beginning with Cycle 3 (21-day cycles) to the end of study (Up to 15 Cycles).
  Interventions: Drug: Alisertib; Drug: Rifampin

INTERVENTIONS:
Drug: Alisertib — Alisertib tablets
  Other Names: MLN8237
Drug: Esomeprazole — Esomeprazole capsules
  Arms: Esomeprazole 40 mg + Alisertib 50 mg
Drug: Rifampin — Rifampin capsules
  Arms: Rifampin 600 mg + Alisertib 50 mg

SUMMARY:
The purpose of this study is to assess the drug-drug interaction (DDI) of either esomeprazole or rifampin on the single-dose PK of alisertib, and to complete an intensive QT study of single and multiple-dose alisertib.

DETAILED DESCRIPTION:
The drug tested in this study is called alisertib. Alisertib is being tested to assess the effect of a proton pump inhibitor and strong metabolic inducer on the PK of a single 50 mg dose of alisertib administered as enteric-coated tablets (ECTs).

The study enrolled 55 patients. Participants received either:

* Esomeprazole 40 mg and Alisertib 50 mg
* Rifampin 600 mg and Alisertib 50 mg

All participants were asked to take one tablet of alisertib either once or twice daily in all cycles. In Cycle 2, participants were asked to take alisertib plus either esomeprazole or rifampin.

This trial was conducted the United States. The overall time to participate in this study was 10 months. Participants made multiple visits to the clinic plus a final visit, 30 days after receiving their last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants 18 years or older
* Histologically or cytologically confirmed metastatic and/or advanced solid tumors or lymphomas
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Expected survival longer than 3 months from enrollment in the study
* Female participants who are post menopausal, surgically sterile, or agree to practice 2 effective methods of contraception or agree to abstain from heterosexual intercourse
* Male participants who agree to practice effective barrier contraception or agree to abstain from heterosexual intercourse

Exclusion Criteria:

* Treatment with any anticancer therapy or any investigational agents within 4 weeks before the first dose of alisertib

  - Known hypersensitivity or intolerance to rifampin (for participants considered for the rifampin drug-drug interaction [DDI] group) or to esomeprazole (for participants considered for the esomeprazole DDI group)
* Recurrent nausea and/or vomiting within 14 days before the first dose of alisertib, and known gastrointestinal (GI) abnormality or GI procedure that could interfere with or modify the oral absorption or tolerance of alisertib
* Participants requiring treatment with clinically significant enzyme inducers within 14 days before the first dose of alisertib and/or requiring the use of these medications during the study
* A medical condition requiring use of pancreatic enzymes; or daily, chronic, or regular use of proton pump inhibitors (PPI); or histamine (H2) receptor antagonists
* Participants requiring systemic anticoagulation (excluding low-dose aspirin, or low-dose anticoagulation to maintain patency of venous access devices).
* Any cardiovascular condition
* Female participants who are lactating or have a positive serum pregnancy test
* Major surgery within the 14 days preceding the first dose of alisertib

  - Life-threatening or uncontrolled medical illness unrelated to cancer
* Newly diagnosed or uncontrolled cancer-related central nervous system (CNS) disease
* Autologous stem cell transplant within 3 months
* Prior allogeneic bone marrow or other organ transplantation

  - Other severe acute or chronic medical or psychiatric condition
* Known or suspected human immunodeficiency virus (HIV) positive or hepatitis B surface antigen-positive status, or known or suspected active hepatitis C infection

Please note there are additional inclusion and exclusion criteria. The study center will determine if you meet all of the criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2013-06-25 (Actual); Primary Completion 2014-08-04 (Actual); Study Completion 2016-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (7):
- United States (7):
  - Sarasota, Florida
  - St Louis, Missouri
  - Oklahoma City, Oklahoma
  - Nashville, Tennessee
  - Dallas, Texas
  - San Antonio, Texas
  - Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 6 investigative sites in the United States from 25 June 2013 to 06 September 2016. Data cut-off for primary analysis was 04 August 2014.
Pre-assignment Details: Participants with a diagnosis of advanced solid tumors or lymphomas were enrolled to receive alisertib 50 mg tablets, orally along with esomeprazole 40 mg, delayed release capsule once daily and alisertib 50 mg along with rifampin 600 mg capsule.
Period: Overall Study
Arm/Group | Esomeprazole 40 mg + Alisertib 50 mg | Rifampin 600 mg + Alisertib 50 mg
Started | 26 | 29
Completed | 18 (Completed=Completed protocol-specified dosing and PK/ECG assessment.) | 19
Not Completed | 8 | 10
Not completed — Didn't complete dosing;PK/ECG assessment | 8 | 10

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Esomeprazole 40 mg + Alisertib 50 mg | Rifampin 600 mg + Alisertib 50 mg | Total
Number analyzed (Participants) | 26 | 29 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (6.90) | 60.4 (10.58) | 61.3 (8.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 21 | 35
  Male | 12 | 8 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 22 | 24 | 46
  Not Reported | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 22 | 26 | 48
  Black or African American | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Asian | 0 | 0 | 0
  American Indian or Alaska Native | 1 | 1 | 2
  Other | 0 | 1 | 1
  Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 29 | 55
Height [Mean (Standard Deviation); unit: cm] | 166.6 (8.90) | 164.8 (9.09) | 165.7 (8.97)
Weight [Mean (Standard Deviation); unit: kg] | 82.07 (20.765) | 77.37 (33.801) | 79.59 (28.242)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index = weight (kg)/ height (m^2).
  kg/m^2 | 29.557 (7.2787) | 28.026 (9.4175) | 28.750 (8.4327)

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Concentration for Alisertib in Presence and Absence of Esomeprazole
Time Frame: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose in Cycle 1 for alisertib without esomeprazole arm; Day 8 pre-dose and at multiple time points (up to 72 hours) post-dose in Cycle 2 for alisertib with esomeprazole arm
Population: The pharmacokinetic (PK) population included participants who completed the protocol-specified dosing and PK sampling requirements in cycle 1 and cycle 2 to have sufficient dosing and plasma concentration-time data to permit calculation of PK parameters.
Measure: Mean (Standard Deviation); unit: nmol/L
Groups:
- Alisertib Without Esomeprazole: Alisertib 50 mg, tablets, orally, once on Day 1 in Cycle 1.
- Alisertib With Esomeprazole: Esomeprazole 40 mg, capsules, orally, once daily on Days 1 to 10 plus alisertib, 50 mg, tablets, orally, once on Day 8, followed by twice daily on Days 11 to 17 in Cycle 2.
Arm/Group | Alisertib Without Esomeprazole | Alisertib With Esomeprazole
Number analyzed (Participants) | 18 | 18
nmol/L | 1542.6 (357.19) | 1804.8 (571.89)
Statistical Analysis 1: Comparison: Alisertib Without Esomeprazole vs Alisertib With Esomeprazole; Test type: Superiority or Other; LS Mean Ratio = 1.14, 90% CI 2-sided [0.97 to 1.35] — Estimates for each PK parameter were obtained using a mixed effects model of log (PK parameter) with fixed terms for the esomeprazole effect and random terms for participants within sequence

2. Primary Outcome: AUClast: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Alisertib in Presence and Absence of Esomeprazole
Time Frame: as for outcome 1
Population: The PK Population included participants who completed the protocol-specified dosing and PK sampling requirements in Cycle 1 and Cycle 2 to have sufficient dosing and plasma concentration-time data to permit calculation of PK parameters.
Measure: Mean (Standard Deviation); unit: hr*nmol/L
Arm/Group | Alisertib Without Esomeprazole | Alisertib With Esomeprazole
Number analyzed (Participants) | 18 | 18
hr*nmol/L | 20427.8 (6813.46) | 25094.4 (5574.04)
Statistical Analysis 1: Comparison: Alisertib Without Esomeprazole vs Alisertib With Esomeprazole; Test type: Superiority or Other; LS Mean Ratio = 1.25, 90% CI 2-sided [1.08 to 1.45] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Alisertib in Presence and Absence of Esomeprazole
Time Frame: as for outcome 1
Population: The PK Population included participants who completed protocol-specified dosing and PK sampling requirements in Cycle 1 and 2 to have sufficient dosing and plasma concentration-time data to permit calculation of PK parameters. Here number of participants analyzed are participants who were evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: hr*nmol/L
Arm/Group | Alisertib Without Esomeprazole | Alisertib With Esomeprazole
Number analyzed (Participants) | 14 | 16
hr*nmol/L | 21371.4 (8138.55) | 26612.5 (6626.40)
Statistical Analysis 1: Comparison: Alisertib Without Esomeprazole vs Alisertib With Esomeprazole; Test type: Superiority or Other; LS Mean Ratio = 1.28, 90% CI 2-sided [1.07 to 1.53] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Alisertib in Presence and Absence of Esomeprazole
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Alisertib Without Esomeprazole | Alisertib With Esomeprazole
Number analyzed (Participants) | 18 | 18
hours | 4.0 [2 to 8] | 3.0 [1 to 8]

5. Primary Outcome: Terminal Phase Elimination Half-life (T1/2) for Alisertib in Presence and Absence of Esomeprazole
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Alisertib Without Esomeprazole | Alisertib With Esomeprazole
Number analyzed (Participants) | 14 | 16
hours | 16.06 (5.398) | 15.96 (5.234)

6. Primary Outcome: Cmax: Maximum Observed Concentration for Alisertib in Presence and Absence of Rifampin
Time Frame: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose in Cycle 1 for alisertib without rifampin arm; Day 8 pre-dose and at multiple time points (up to 72 hours) post-dose in Cycle 2 for alisertib with rifampin arm
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nmol/L
Groups:
- Alisertib Without Rifampin: Alisertib 50 mg, tablets, orally, once on Day 1 in Cycle 1.
- Alisertib With Rifampin: Rifampin 600 mg, capsules, orally, once daily on Days 1 to 10 plus alisertib, 50 mg, tablets, orally, once on Day 8, followed by twice daily on up Days 11 to 17 in Cycle 2.
Arm/Group | Alisertib Without Rifampin | Alisertib With Rifampin
Number analyzed (Participants) | 20 | 20
nmol/L | 1561.4 (661.81) | 1581.5 (519.68)
Statistical Analysis 1: Comparison: Alisertib Without Rifampin vs Alisertib With Rifampin; Test type: Superiority or Other; LS Mean Ratio = 1.03, 90% CI 2-sided [0.84 to 1.26] — [estimate comment as in outcome 1, analysis 1]

7. Primary Outcome: AUC(Last): Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Alisertib in Presence and Absence of Rifampin
Time Frame: as for outcome 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr*nmol/L
Arm/Group | Alisertib Without Rifampin | Alisertib With Rifampin
Number analyzed (Participants) | 20 | 20
hr*nmol/L | 19732.0 (8489.24) | 9470.5 (2653.60)
Statistical Analysis 1: Comparison: Alisertib Without Rifampin vs Alisertib With Rifampin; Test type: Superiority or Other; LS Mean Ratio = 0.51, 90% CI 2-sided [0.41 to 0.62] — [estimate comment as in outcome 1, analysis 1]

8. Primary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Alisertib in Presence or Absence of Rifampin
Time Frame: as for outcome 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr*nmol/L
Arm/Group | Alisertib Without Rifampin | Alisertib With Rifampin
Number analyzed (Participants) | 12 | 8
hr*nmol/L | 17258.3 (6163.60) | 8955.0 (2389.25)
Statistical Analysis 1: Comparison: Alisertib Without Rifampin vs Alisertib With Rifampin; Test type: Superiority or Other; LS Mean Ratio = 0.53, 90% CI 2-sided [0.41 to 0.70] — [estimate comment as in outcome 1, analysis 1]

9. Primary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Alisertib in Presence and Absence of Rifampin
Time Frame: as for outcome 6
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Alisertib Without Rifampin | Alisertib With Rifampin
Number analyzed (Participants) | 20 | 20
hours | 4.0 [1 to 23] | 2.1 [1 to 6]

10. Primary Outcome: Phase Elimination Half-life (T1/2) for Alisertib in Presence and Absence of Rifampin
Time Frame: as for outcome 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Alisertib Without Rifampin | Alisertib With Rifampin
Number analyzed (Participants) | 12 | 8
hours | 16.30 (6.608) | 8.17 (5.476)

11. Primary Outcome: Change From the Time-matched Baseline in the Individually Corrected QTc Interval (QTcI)
Time Frame: Baseline, Days 1 and 10 multiple timepoints postdose (up to 24 hours) in Cycle 1
Population: The electrocardiogram (ECG) QTc population included participants who received at least 1 dose of alisertib and have at least 1 post-baseline ECG.
Measure: Mean (95% Confidence Interval); unit: milliseconds (msec)
Groups:
- Alisertib: Alisertib 50 mg, tablets, orally, once on Day 1, followed by twice daily on Days 4 to 10, followed by a 14-day rest period in Cycle 1.
Arm/Group | Alisertib
Number analyzed (Participants) | 55
milliseconds (msec)
  Day 10, 0 hour postdose | -2.2 [NA to 0.99] — One sided 95% Upper Confidence Bounds was estimated.
  Day 1, 0.5 hour postdose | -3.7 [NA to -1.63] — One sided 95% Upper Confidence Bounds was estimated.
  Day 10, 0.5 hour postdose | -5.4 [NA to -2.24] — One sided 95% Upper Confidence Bounds was estimated.
  Day 1, 1 hour postdose | -4.5 [NA to -2.37] — One sided 95% Upper Confidence Bounds was estimated.
  Day 10, 1 hour postdose | -3.5 [NA to -0.4] — One sided 95% Upper Confidence Bounds was estimated.
  Day 1, 2 hours postdose | -4.0 [NA to -1.94] — One sided 95% Upper Confidence Bounds was estimated.
  Day 10, 2 hours postdose | -1.6 [NA to 1.54] — One sided 95% Upper Confidence Bounds was estimated.
  Day 1, 3 hours postdose | -2.5 [NA to -0.42] — One sided 95% Upper Confidence Bounds was estimated.
  Day 10, 3 hours postdose | -2.3 [NA to 0.89] — One sided 95% Upper Confidence Bounds was estimated.
  Day 1, 4 hours postdose | -1.2 [NA to 0.9] — One sided 95% Upper Confidence Bounds was estimated.
  Day 10, 4 hours postdose | -1.2 [NA to 1.91] — One sided 95% Upper Confidence Bounds was estimated.
  Day 1, 6 hours postdose | -0.9 [NA to 1.15] — One sided 95% Upper Confidence Bounds was estimated.
  Day 10, 6 hours postdose | -3.5 [NA to -0.33] — One sided 95% Upper Confidence Bounds was estimated.
  Day 1, 8 hours postdose | -0.5 [NA to 1.61] — One sided 95% Upper Confidence Bounds was estimated.
  Day 10, 8 hours postdose | -0.4 [NA to 2.75] — One sided 95% Upper Confidence Bounds was estimated.
  Day 1, 10 hours postdose | -1.5 [NA to 0.56] — One sided 95% Upper Confidence Bounds was estimated.
  Day 10, 10 hours postdose | -2.4 [NA to 0.73] — One sided 95% Upper Confidence Bounds was estimated.
  Day 1, 24 hours postdose | -3.3 [NA to -1.2] — One sided 95% Upper Confidence Bounds was estimated.

12. Secondary Outcome: Change From the Time-matched Baseline in the Fridericia Correction of QTc (QTcF)
Time Frame: Baseline, Days 1 and 10 multiple timepoints postdose (up to 24 hours) in Cycle 1
Population: as for outcome 11
Measure: Mean (95% Confidence Interval); unit: milliseconds (msec)
Arm/Group | Alisertib
Number analyzed (Participants) | 55
milliseconds (msec)
  Day 10, 0 hour postdose | -2.4 [NA to 0.7] — One sided 95% Upper Confidence Bounds was estimated.
  Day 1, 0.5 hour postdose | -3.9 [NA to -1.8] — One sided 95% Upper Confidence Bounds was estimated.
  Day 10, 0.5 hour postdose | -5.3 [NA to -2.19] — One sided 95% Upper Confidence Bounds was estimated.
  Day 1, 1 hour postdose | -4.6 [NA to -2.54] — One sided 95% Upper Confidence Bounds was estimated.
  Day 10, 1 hour postdose | -3.9 [NA to -0.76] — One sided 95% Upper Confidence Bounds was estimated.
  Day 1, 2 hours postdose | -3.5 [NA to -1.51] — One sided 95% Upper Confidence Bounds was estimated.
  Day 10, 2 hours postdose | -2.5 [NA to 0.63] — One sided 95% Upper Confidence Bounds was estimated.
  Day 1, 3 hours postdose | -2.1 [NA to -0.09] — One sided 95% Upper Confidence Bounds was estimated.
  Day 10, 3 hours postdose | -2.6 [NA to 0.55] — One sided 95% Upper Confidence Bounds was estimated.
  Day 1, 4 hours postdose | 0 [NA to 2.07] — One sided 95% Upper Confidence Bounds was estimated.
  Day 10, 4 hours postdose | -1.3 [NA to 1.87] — One sided 95% Upper Confidence Bounds was estimated.
  Day 1, 6 hours postdose | -0.5 [NA to 1.5] — One sided 95% Upper Confidence Bounds was estimated.
  Day 10, 6 hours postdose | -4.1 [NA to -0.92] — One sided 95% Upper Confidence Bounds was estimated.
  Day 1, 8 hours postdose | 0 [NA to 2.1] — One sided 95% Upper Confidence Bounds was estimated.
  Day 10, 8 hours postdose | -1.6 [NA to 1.54] — One sided 95% Upper Confidence Bounds was estimated.
  Day 1, 10 hours postdose | -1.2 [NA to 0.9] — One sided 95% Upper Confidence Bounds was estimated.
  Day 10, 10 hours postdose | -3.5 [NA to -0.3] — One sided 95% Upper Confidence Bounds was estimated.
  Day 1, 24 hours postdose | -3.8 [NA to -1.72] — One sided 95% Upper Confidence Bounds was estimated.

13. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A Serious Adverse Event (SAE) A serious is any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.
Time Frame: From the first dose through 30 days after administration of the last dose of study drug (up to 328 days)
Population: The safety population included all participants who received at least 1 dose of alisertib. According to the protocol analysis planned, primary purpose of the study was to observe the drug-drug interaction of either esomeprazole or rifampin on the single-dose of alisertib.
Measure: Number; unit: participants
Arm/Group | Esomeprazole 40 mg + Alisertib 50 mg | Rifampin 600 mg + Alisertib 50 mg
Number analyzed (Participants) | 26 | 29
participants
  AEs | 25 | 27
  SAEs | 9 | 11

ADVERSE EVENTS:
Time Frame: From the first dose through 30 days after administration of the last dose of study drug (up to 328 days)
Description: Any AE spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. According to the protocol analysis planned, primary purpose of the study was to observe the drug-drug interaction of either esomeprazole or rifampin on the single-dose of alisertib.
Arm/Group | Esomeprazole 40 mg + Alisertib 50 mg | Rifampin 600 mg + Alisertib 50 mg
All-Cause Mortality (participants affected / at risk) | 1/26 | 3/29
Serious Adverse Events (participants affected / at risk) | 9/26 | 11/29
Other Adverse Events (participants affected / at risk) | 25/26 | 25/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Esomeprazole 40 mg + Alisertib 50 mg (N=26) | Rifampin 600 mg + Alisertib 50 mg (N=29)
Vomiting (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 — One treatment-emergent death occurred during treatment with rifampin and alisertib and is not related.
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — One treatment-emergent death occurred during treatment with esomeprazole and alisertib and is not related.
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 — One treatment-emergent death occurred during treatment with rifampin and alisertib and is not related.
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 2
Orthostatic hypotension (Vascular disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 — One treatment-emergent death occurred during treatment with rifampin and alisertib and is not related.
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Esomeprazole 40 mg + Alisertib 50 mg (N=26) | Rifampin 600 mg + Alisertib 50 mg (N=29)
Diarrhoea (Gastrointestinal disorders) | 15 | 4
Stomatitis (Gastrointestinal disorders) | 11 | 6
Vomiting (Gastrointestinal disorders) | 7 | 5
Nausea (Gastrointestinal disorders) | 7 | 4
Abdominal pain (Gastrointestinal disorders) | 4 | 5
Constipation (Gastrointestinal disorders) | 4 | 1
Dry mouth (Gastrointestinal disorders) | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 1
Fatigue (General disorders) | 12 | 10
Oedema peripheral (General disorders) | 2 | 3
Asthenia (General disorders) | 3 | 0
Pyrexia (General disorders) | 2 | 1
Non-cardiac chest pain (General disorders) | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 14 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Rash macular (Skin and subcutaneous tissue disorders) | 3 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 10 | 7
Anaemia (Blood and lymphatic system disorders) | 7 | 8
Leukopenia (Blood and lymphatic system disorders) | 4 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 4
Lymphopenia (Blood and lymphatic system disorders) | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 7 | 3
Dehydration (Metabolism and nutrition disorders) | 4 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Gamma-glutamyltransferase increased (Investigations) | 3 | 4
Alanine aminotransferase increased (Investigations) | 3 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 2
Weight decreased (Investigations) | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dizziness (Nervous system disorders) | 3 | 1
Headache (Nervous system disorders) | 2 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 0
Urinary tract infection (Infections and infestations) | 1 | 2
Vision blurred (Eye disorders) | 2 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.